CLINICAL TRIAL: NCT05001867
Title: Comparing Conventional Abdominal Ultrasound Scanning Versus a Robotic Assisted Ultrasonography System (ROBUST): a Pilot Study
Brief Title: Comparing Conventional Abdominal Ultrasound Scanning Versus a Robotic Assisted Ultrasonography System (ROBUST)
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Collaborators: Sengkang General Hospital (Other); Servo Dynamics (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2017/3049
Record Dates: First submitted 2021-07-25; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Work-related Musculoskeletal Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Work-related musculoskeletal disorders (WRMSD) among sonographers/radiographers are prevalent in the healthcare industry. This pilot study will evaluate the use of a robotic assisted ultrasonography system (ROBUST) against the conventional abdominal ultrasound scanning procedure. The ROBUST will be developed to provide 6 degrees of freedom to allow radiographers to perform abdominal scanning without having to reach over patients.

10 sonographers with at least 5 years of experience will be recruited from SGH and SKH, to perform abdominal ultrasound scans on healthy volunteers. Each sonographer will be randomly assigned to scan a volunteer using conventional abdominal ultrasound scanning procedure and with ROBUST respectively. The study will be done in 2 phases, separated by at least a 1-month interval between scans.

Phase 1: Scanning of volunteer using conventional abdominal ultrasound scanning procedure.

Phase 2: Scanning of volunteer using ROBUST. Outcome measures will include ultrasound image quality, sonographer feedback and comfort level as well as satisfaction feedback from healthy volunteers. A panel of 4 reviewers, consisting of 2 radiologists and 2 senior radiographers will be invited to grade the images, using a 3-point Likert scale. The duration of each scanning will be recorded. The comfort level reported by sonographers will be assessed using the SGH Comfort Level Survey. In addition, the comfort level of healthy volunteers will also be assessed using a satisfaction questionnaire.

DETAILED DESCRIPTION:
* 10 participating sonographers will be recruited from SGH and SKH to perform abdominal ultrasound scanning.
* 10 healthy volunteers of average body habitus with BMI <30, abdominal circumference <102cm will be recruited.
* Each sonographer will be randomly assigned to scan 1 healthy volunteer. The same volunteer will be scanned twice with an interval of at least 1 month between two scans: once using conventional abdominal ultrasound scanning procedure and once using ROBUST.
* During the session, markers coated with a retroreflective material to reflect light to the motion capture camera will be pasted on participating sonographers on various parts of the upper limb.
* Surface electromyography (sEMG) electrodes will be affixed on sonographers' upper trapezius, deltoid, biceps, triceps, wrist extensors and flexors to monitor muscle activities.
* The healthy volunteer will lie on a plinth with the participating sonographer seated next to him/her. The sonographer will then perform scanning on various abdominal organs following the point of reference and scanning approach as indicated.
* The same ultrasound scanner and probe type will be used on all volunteers by all sonographers.
* Static bilateral grip strength of participating sonographers will be measured using a dynamometer before and after each scan.
* At the end of both scans, participating sonographers will be required to complete a survey on comfort level.
* At the end of both scans, healthy volunteers will be required to complete a survey on satisfaction level.
* The quality of the images from both scans will be rated by 4 readers: 2 consultant radiologists and 2 senior radiographers. A photometer will be used to ensure all readers interpret images directly from a designated monitor under consistent lighting condition.

ELIGIBILITY:
Inclusion Criteria:

Sonographer:

-Experienced sonographers/ radiographers with more than 5 years of experience

Healthy volunteer:

* Inclusion criteria: - BMI <30
* Abdominal circumference <102cm

Exclusion Criteria:

Sonographer:

-Participating sonographers with previously reported work-related or non-work related musculoskeletal discomfort or injury

Healthy volunteer:

-Pregnancy

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 sonographers from SGH or SKH and 10 healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Comparison of quality of ultrasound image for manual scanning and robot scanning | During the scan
Kinematic data, Range of Motion from motion capture system | During the scan
Muscle activation from EMG data | During the scan
Static bilateral grip strength | Immediately before the scan and immediately after the scan
Questionnaire on comfort level from sonographers | immediately after the scan
Questionnaire on Satisfaction level from healthy volunteers | immediately after the scan

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Sengkang General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No